CLINICAL TRIAL: NCT00491855
Title: Phase I Trial of Intraperitoneal Oxaliplatin and Paclitaxel Plus Intravenous Paclitaxel and Bevacizumab in the Treatment of Advanced Peritoneal Carcinomatosis
Brief Title: Oxaliplatin and Paclitaxel Plus Bevacizumab in Advanced Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1068
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Peritoneal Cancer
Keywords: Advanced Peritoneal Carcinomatosis; Peritoneal Cancer; Bevacizumab; Avastin; vascular endothelial growth factor; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Oxaliplatin; Eloxatin; Paclitaxel; Taxol
MeSH Terms: interventions — Bevacizumab; Oxaliplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Oxaliplatin + Paclitaxel (Experimental): One cycle of treatment is 21 days. Bevacizumab starting dose level 2.5 mg/kg given intravenously on day 1. Oxaliplatin starting dose level 25 mg/m^2 given intraperitoneally on day 2. Paclitaxel starting dose level 110 mg/m^2 given continuous infusion on day 1 and 30 mg/m^2 given intraperitoneally on day 8.
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Starting dose level 2.5 mg/kg given intravenously on day 1.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Oxaliplatin — Starting dose level 25 mg/m^2 given intraperitoneally on day 2.
  Other Names: Eloxatin
Drug: Paclitaxel — Starting dose level 110 mg/m^2 given continuous infusion on day 1 and 30 mg/m^2 given intraperitoneally on day 8.
  Other Names: Taxol

SUMMARY:
The goal of this clinical research is to learn acceptable dosages of paclitaxel, oxaliplatin, and Avastin (bevacizumab) that can be given in combination to patients with advanced peritoneal carcinomatosis. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Paclitaxel is designed to block cancer cells from dividing, which may cause them to die.

Oxaliplatin is designed to keep new cancer cells from growing

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Study Drug Dose Levels:

Up to 12 study drug dose levels will be tested in this study. Participants will be enrolled in groups of 3. The first 3 participants will be enrolled at the lowest dose level. If there are no intolerable side effect seen, the next 3 participants will be enrolled into the next higher dose level. This will continue until acceptable dose levels of the study drugs are found. The dose level that you are assigned to will depend on when you enroll on this study. You will receive the same dose level for the entire study unless you develop side effects, in which case doses of the drugs will be decreased by your doctor.

Drug Administration:

If you agree to participate in this study, you will have a catheter placed in your abdomen before receiving study drug. A catheter is a sterile flexible tube that will be placed while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

On Day 1, you will receive bevacizumab followed by paclitaxel through a needle in your vein over 24 hours.

On Day 2, after you have completed the paclitaxel infusion, you will be given about 1 quart of fluid containing oxaliplatin into the abdomen through the catheter over 15 minutes.

On Day 8, you will be given about 1 quart of fluid containing paclitaxel into the abdomen through the catheter over 15 minutes.

Every 21 days is called a study "cycle."

Study Visits:

During each cycle, you will see your doctor in his office to make sure that you are still eligible to receive study drugs.

* Blood (about 1 tablespoon) will be drawn for routine tests each day during hospitalization and then once a week as an outpatient.
* A urine sample will be collected once each cycle for routine tests.
* You will have scans such as a chest x-ray, CT, MRI, Positron emission tomography (PET), and/or PET/CT scan after every 2 cycles (6 weeks) or earlier if the study doctor thinks it is in your best interest, or the cancer gets worse. These scans are to check the status of the disease. If the study doctor thinks it is more appropriate for you, other types of scans may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form.

Length of Study:

You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

If you are taken off study, you will be asked to have an end-of-study visit. At this visit, the following tests will be performed:

* Blood (about 1 tablespoon) and urine will be collected for routine tests.
* You will have repeat scans such as a chest x-ray, CT, MRI, PET, and/or PET/CT scan to check the status of the disease. If the study doctor thinks it is more appropriate for you, other types of scans may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form.

This is an investigational study. Paclitaxel, oxaliplatin, and bevacizumab are FDA-approved drugs, but their use in this study is investigational. Up to 72 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have advanced peritoneal carcinomatosis: they have either a disease where there is no established standard of care therapy or have failed one or more prior therapy. These include, but not limited to, recurrent epithelial ovarian cancer, advanced endometrial cancer, advanced gastric cancer, advanced colorectal cancer, and advanced primary peritoneal mesothelioma without significant chest involvement. Previous intraperitoneal therapy with different agents is allowed as long as their diseases have progressed.
2. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status < or = 2 (0-2).
3. Patients must have normal organ and marrow function as defined below: Absolute neutrophil count > or = 1,500/mcL Platelets > or = 100,000/mcL Total bilirubin < or = 2.0 and alanine aminotransferase (ALT) <2.5 * the institutional upper limit of normal; Creatinine < or = 2.0 mg/dL or creatinine clearance > or = 40mL/min/1.73m2.
4. Patients must be able to understand and the willingness to sign an Institutional Review Board (IRB)-approved written informed consent document.
5. Patients must have evidence of peritoneal carcinomatosis that is evaluable by computer tomography (CT) or magnetic resonance imaging (MRI).
6. In the clinical judgment of the investigator, patients must have adequate potential intraperitoneal fluid distribution with no gross fluid loculations and adhesions that would significantly affect intraperitoneal drug distribution. This determination may be made based on documented clinical, imaging or laboratory assessment.
7. Patients must have prothrombin time (PT)/ partial thromboplastin time (PTT) within 1.2 * the institutional upper limit of normal or < 3 * the institutional upper limit of normal on anticoagulants.
8. Patients must have resting blood pressure no greater than 140 mmHg(systolic) or 90 mmHg (diastolic) for eligibility. Initiation or adjustment of blood pressure medication is permitted prior to study entry.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, symptomatic cardiac arrhythmia, active bleeding, active thrombosis, or psychiatric illness/social situations that would limit compliance with study requirements.
2. History of allergic reactions to the study drugs or their analogs.
3. Failure to recover from any prior surgery within 4 weeks of study entry.
4. Pregnant or lactating. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry, for the duration of study participation and for at least 3 months after the last treatment.
5. Any treatment specific for tumor control within 3 weeks of study drugs; or within 2 weeks if cytotoxic agents were given weekly (within 6 wks for nitrosoureas or mitomycin C), or within 5 half-lives for target agents with half lives and pharmacodynamic effects lasting less than 5 days (that include but are not limited to erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents); or failure to recover from the toxic effect of any therapy prior to study entry.
6. Serious non-healing wound, ulcer, bone fracture (including abdominal fistula, gastrointestinal perforation or intra-abdominal abscess), or history of bleeding diathesis.
7. History of radiotherapy to the abdominal and pelvic regions or history of multiple abdominal surgeries that contraindicates this protocol therapy.
8. Urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
9. Grade 2 or greater neuropathy, and history of brain or leptomeningeal metastases that significantly increase risks of intracranial bleeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continual assessment during each 21 day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org